CLINICAL TRIAL: NCT06012630
Title: Ultrasound Evaluation of the Median Nerve in Patients With Rheumatoid Arthritis and Its Relationship With Disease Activity
Brief Title: Carpal Tunnel Syndrome Evaluation With Ultrasound in Rheumatoid Arthritis Patients
Status: Completed | Type: Observational
Sponsor: Burak Tayyip Dede (Other Government)
Responsible Party: Sponsor-Investigator, Burak Tayyip Dede, Physical Medicine and Rehabilitation, Istanbul Training and Research Hospital
Organization: Istanbul Training and Research Hospital (Other Government)
Other Study IDs: 22/04/2022; 2011-KAEK-50;126
Record Dates: First submitted 2023-08-17; First posted 2023-08-25 (Actual); Last update posted 2023-08-25 (Actual); Status verified 2023-08

CONDITIONS: Median Nerve Entrapment
Keywords: Rheumatoid arthritis; Ultrasound; Carpal Tunnel Syndrome
MeSH Terms: conditions — Median Neuropathy; Arthritis, Rheumatoid; Carpal Tunnel Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 8 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- group 1: RA without CTS: Rheumatoid arthritis patients without a diagnosis of CTS based on clinical findings and physical examination
  Interventions: Diagnostic Test: Ultarsound
- group 2: RA with CTS: Rheumatoid arthritis patients with a diagnosis of CTS based on clinical findings and physical examination
  Interventions: Diagnostic Test: Ultarsound
- group:3 Healthy Control: Healthy Control without rheumatologic disease and Carpal tunnel syndrome
  Interventions: Diagnostic Test: Ultarsound

INTERVENTIONS:
Diagnostic Test: Ultarsound — Median nerve evaluation of participants with ultrasound

SUMMARY:
In rheumatoid arthritis (RA) patients, the diagnosis of Carpal tunnel syndrome (CTS) was made based on clinical findings and physical examinations. Then, the cross-sectional areas of the participants' median nerves from different levels were measured. Meidolateral and anteroposterior diameter were measured at the level of the carpal tunnel inlet. Flattening ratio was calculated. wrist to forearm ratio and wrist to forearm difference were calculated. The obtained data were compared between RA with CTS, RA without CTS and healthy control.

ELIGIBILITY:
Inclusion Criteria:

* RA patients identified according to the 2010 American College of Rheumatology/Europan Leage Against Rheumatism classification criteria
* healthy controls (HC) with no history of rheumatic diseases and CTS.
* Individuals aged 18-65 years.

Exclusion Criteria:

* thoese with hypothyroidism,
* gout,
* diabetes mellitus,
* history of CTS surgery,
* upper extremity plexopathy,
* polinöropathy,
* uncontrollable fibromyalgia,
* steroid injection for CTS
* For the HC group, those with phalen or tinnel detected in at least one wrist and those with bifid median nerve detected during US evaluation were not included in the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: RA patients identified according to the 2010 American College of Rheumatology/Europan Leage Against Rheumatism classification criteria healthy controls (HC) with no history of rheumatic diseases and CTS.
Sampling Method: Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2023-01-15 (Actual); Primary Completion 2023-07-01 (Actual); Study Completion 2023-08-15 (Actual)

PRIMARY OUTCOMES:
Comparison of US findings among participants | 6 months
  Comparison of US findings among participants

SECONDARY OUTCOMES:
Relationship between US findings and disease activity in the patient group | 6 months
  The correlation between the US findings of the participants in the patient group and the CDA, which evaluates disease activity, was examined.

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul Training and Resarch Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes